CLINICAL TRIAL: NCT01014663
Title: Comparison of Non-contact Boxing Training and Traditional Therapeutic Exercise on Functional Outcomes in Persons With Parkinson's Disease
Brief Title: Non-contact Boxing Training and Traditional Therapeutic Exercise for Persons With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Indianapolis (Other)
Responsible Party: Principal Investigator, Stephanie Miller, Associate Professor, University of Indianapolis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXB-01
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; exercise; training program; rehabilitation; boxing
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic Exercise (Active Comparator)
  Interventions: Behavioral: Traditional Therapeutic Exercise
- Non-Contact Boxing Training (Active Comparator)
  Interventions: Behavioral: Non-Contact Boxing Training

INTERVENTIONS:
Behavioral: Traditional Therapeutic Exercise — The therapeutic exercise program will consist of warm-up and stretching, seated and standing range of motion activities, endurance and resistance training, balance training and a cool down. Training will take place for 36 sessions, three times/week for 60-90 minutes per session.
  Arms: Therapeutic Exercise
Behavioral: Non-Contact Boxing Training — Non-contact boxing training will consist of warm-up and stretching, non-contact boxing training (including punching a focus mitt, speed and heavy punching bags), endurance training activities, strength and resistance training, and a cool down. Training will take place for 36 sessions, three times/week for 60-90 minutes per session.
  Arms: Non-Contact Boxing Training

SUMMARY:
The primary purpose of this study is to compare the effects of a non-traditional boxing training program to a traditional therapeutic exercise program on activity and participation outcomes in persons with Parkinson's disease. Thirty participants will be randomly assigned to participate in either non-contact boxing training or traditional therapeutic exercise for 36 sessions over 12 weeks. Participants will be measured immediately before (pre-test) and after (post-test) the intervention.

DETAILED DESCRIPTION:
Physical therapists commonly treat patients with Parkinson's disease. Typical clinical interventions used by physical therapists including strengthening, stretching and aerobic training have been shown to improve function and quality of life of persons with Parkinson's disease. Alternative exercise interventions that incorporate non-traditional concepts, such as tango dance, tai chi and taiji have also been found to lead to improvements in function in persons with Parkinson's disease. It is important that comparisons between different types of exercise programs for persons with Parkinson's disease be explored in order to determine effective options for care.

Here in Indianapolis, Indiana, individuals with Parkinson's disease have a unique opportunity for alternative exercise with the recent development of the popular non-contact boxing training program offered by the Rock Steady Boxing Foundation. Therefore, the purpose of this study is to compare the effects of the non-traditional boxing training program to a traditional therapeutic exercise program on activity and participation outcomes in persons with Parkinson's disease.

Thirty participants with Parkinson's disease will be recruited from Central Indiana. All potential participants will be screened to determine eligibility for the study. Participants who are eligible and give consent will be randomly assigned to participate in either the non-contact boxing training or the traditional therapeutic exercise program for 36 sessions lasting over 12 weeks with 60-90 minutes of exercise each session. Participants will be measured immediately before (pre-test) and after (post-test) the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's disease
* currently not receiving physical therapy services
* medically stable with a physician release stating approval to enter an exercise program
* independently ambulatory in the home setting with or without the use of an assistive device
* able to follow at least three step verbal commands
* available for the entire period of the study
* have transportation to and from training and measurement sessions

Exclusion Criteria:

* preexisting neurological conditions other than Parkinson's disease
* current musculoskeletal conditions that would limit participation in either training program
* significant orthopedic surgery within the past six months
* past brain surgery or brain stimulator implant
* currently known pregnant
* pre-existing cardiovascular conditioner that would prohibit participation in an exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Mobility: Measured with the Timed Up and Go Test; Four-Square Step Test; Six-Minute Walk Test; Berg Balance Scale; Functional Reach Test | Each outcome measures is assessed at pre-test (immediately before intervention), post-test (immediately after the 12 week intervention).

SECONDARY OUTCOMES:
Participation: measured with the Activities Specific Balance Confidence Scale and the Parkinson's disease Quality of Life Scale | Each outcome measures is assessed at pre-test (immediately before intervention), post-test (immediately after the 12 week intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Combs, PT, PhD, NCS, Principal Investigator — University of Indianapolis; Dyer M Diehl, PT, PhD, Principal Investigator — University of Indianapolis; William H Staples, PT, DPT, GCS, Principal Investigator — University of Indianapolis
Locations (1):
- University of Indianapolis, Krannert School of Physical Therapy, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886